CLINICAL TRIAL: NCT06571448
Title: A Phase 2 Randomized, Double-blind and Placebo-controlled Study to Assess the Efficacy, Safety, and Tolerability of SR750 in Patients With Trigeminal Neuralgia
Brief Title: Efficacy, Safety, and Tolerability of SR750 in Patients With Trigeminal Neuralgia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai SIMR Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SR750-202
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Trigeminal Neuralgia
Keywords: Trigeminal Neuralgia; SR750
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SR750 high dose (Experimental)
  Interventions: Drug: SR750 tablet
- SR750 low dose (Experimental)
  Interventions: Drug: SR750 tablet
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SR750 tablet — SR750 high dose BID orally for 6 weeks
  Arms: SR750 high dose
Drug: SR750 tablet — SR750 low dose BID orally for 6 weeks
  Arms: SR750 low dose
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy，safety and tolerability of SR750 in patients with trigeminal neuralgia (TN). Patients will receive SR750 (study drug) or placebo for 6 weeks and keep a diary of daily pain. The study duration for each patient is up to 11 weeks.

DETAILED DESCRIPTION:
This is a phase 2, randomized, double-blind study comparing SR750 with placebo in patients with trigeminal neuralgia. It consists of a screening period, a double-blind treatment period, and a post-treatment safety follow-up period. Baseline pain intensity and number of paroxysms will be taken in the run-in period of screening period and will be checked for eligibility. Around 162 eligible subjects will be recruited and randomized into three arms at 1:1:1 ratio to receive SR750 high dose twice a day (BID) , SR750 low dose BID or placebo BID for 6 weeks. Subjects, investigators, all clinical study site staffs, and the Sponsor will remain blinded to treatment assignment during the study. Subjects will be asked to record the number of paroxysms of pain, severity of daily average pain of paroxysms and severity of daily worst pain in e-diary over the last 24 hours every night before going to bed. After completion of double-blind period, subjects will continue to complete the safety follow-up.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of trigeminal neuralgia as per International Classification of Headache Disorders third version (ICHD-3) criteria
* Subjects must have completed at least 5 daily pain score and experienced ≥3 paroxysms per day with a daily average pain sore of ≥4 on PI-NRS during the five days prior to randomization.
* Willing and able to undergo washout of prohibited medication as per protocol requirements and refrain from use of the prohibited medication throughout the study period.
* Female subjects must be non-pregnant and non-lactating.

Key Exclusion Criteria:

* Secondary trigeminal neuralgia
* Painful trigeminal neuropathies
* Other pains that cannot be clearly differentiated from the pain associated with TN or may interfere with the pain assessment
* Subjects have previously undergone microvascular decompression (MVD), sensory rhizotomy of trigeminal nerve, radiofrequency ablation (RFA), percutaneous balloon compression (PBC), permanent lesion of trigeminal semilunar ganglion, botulinum toxin type A for the treatment of TN within 6 months prior to screening. Subjects with severe complication after therapeutic procedure would also be excluded.
* Known history of human immunodeficiency virus (HIV) or active infection of hepatitis B virus (HBV), hepatitis C virus (HCV) or Treponema Pallidum

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Daily Average Pain Score (DAPS) | up to week 6
  Change from baseline to week 6 in the weekly average of the daily average pain score (DAPS) of paroxysms using pain intensity numerical rating scale (PI-NRS).The PI-NRS consists of an 11-point numeric scale ranging from 0 (no pain) to 10 (worst imaginable pain). Participants described their pain during the past 24 hours by choosing the appropriate number between 0 and 10.

SECONDARY OUTCOMES:
Proportion of responders | up to week 6
  Proportion of subjects who meets one of the following criteria,
  * Patient Global Impression of Change (PGIC) response of "Much Improved" or "Very Much Improved" at Week 6. Subjects will select a value to represent their overall status since the start of the study on a 7-point scale of PGIC on which 1 corresponds to "very much improved", 2 corresponds to "much improved", 3 corresponds to "slightly improved" 4 corresponds to "no change", 5 corresponds to "slightly worse", 6 corresponds to "much worse", and 7 corresponds to "very much worse".
  * A reduction of ≥2 points from baseline in mean pain score at Week 6
  * A reduction of ≥30% from baseline in mean pain score at Week 6
  * A reduction of ≥50% from baseline in mean pain score at Week 6
  * A reduction of ≥30% from baseline in mean number of paroxysms at Week 6
  * A reduction of ≥50% from baseline in mean number of paroxysms at Week 6
  * A reduction of ≥30% from baseline in mean worst pain score at Week 6
Mean pain score by week | up to week 6
  Change from baseline in weekly mean pain score. The daily pain score will be measured by PI-NRS described as above.
Mean worst pain score by week | up to week 6
  Change from baseline in mean worst pain score by week. The daily worst pain score will be measured by PI-NRS described as above.
Mean number of paroxysms by week | up to week 6
  Change from baseline in mean number of paroxysms by week
Mean continuous pain score by week | up to week 6
  Change from baseline in mean continuous pain score by week. The daily continuous pain score will be measured by PI-NRS described as above.
Proportion of subjects with continuous pain at week 6 | up to week 6
  Change of proportion from baseline
Hospital Anxiety and Depression Scale (HADS) | up to week 6
  Change of HADS from baseline. The HADS is a self-administered questionnaire consisting of two subscales, one for anxiety (HADS-A Subscale) and the other for depression (HADS-D Subscale). Each subscale consists of 7 items, and subjects will rate each item as it applies to them 0 points = absence of anxiety or depression; 3 points = severe anxiety or depression. The HADS-A Subscale analyzes generalized anxiety states, including anxious feelings, restlessness, anxious thoughts, and panic attacks. The HADS-D Subscale focuses on states of loss of interest and reduced pleasure response (reduced enjoyment mood). Each subscale will receive a score from 0 to 21, with bigger number indicating more severe symptom.
Use of rescue medication | up to week 7
  Including the first time to use rescue medication, total amount and proportion

OTHER OUTCOMES:
Adverse events | up to week 7
  To collect the adverse events during the study
Plasma concentration of SR750 and its metabolite | up to day 43
  To measure the plasma concentration of SR750 and its metabolite after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bifa Fan, MD, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No